CLINICAL TRIAL: NCT04796181
Title: Single Center, Single Blinded, Prospective Validation Study for the Accuracy and Safety Evaluation of Neteera 130H, a Novel, Radar-based Contact-free Device for Heart and Respiratory Rate Measurements
Brief Title: Heart Rate and Respiratory Rate Measurements by a Novel, Radar-based Device
Status: Completed | Type: Observational
Sponsor: Neteera Technologies Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: NET-MED-002-EXT
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-02

CONDITIONS: Healthy Subjects; Chronic Conditions, Multiple
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Neteera 130H — The Neteera 130H will used to perform measurements in proximity to study participants.

SUMMARY:
A single center, single blinded, prospective validation (including extension0 study for the accuracy and safety evaluation of Neteera 130H, a novel, radar-based contact-free device for heart and respiratory rate measurements.

DETAILED DESCRIPTION:
This is a single-blinded, prospective validation study for the accuracy and safety evaluation of Neteera 130H, a novel, radar-based contact-free device for heart and respiratory rate measurements compared to reference devices.

Each subject will have a single study visit in which the subjects will be screened and upon eligibility confirmation, will undergo HR and RR measurements using the investigational device as well as the reference devices. In a previous clinical trial (NET-MED-002) 100 subjects were measured in the sitting position. In the extension study part (NET-MED-002-EXT), 70 eligible subjects, 18 years old and above, suffering from chronic medical conditions, will be enrolled. In this extension part, 70 of the subjects will be measured while randomly assigned into one of two groups - 35 subjects in group A (sitting position) and 35 subjects in sleep posture//group B (lying in bed/sleeping posture position) in a ratio of 1:1. Data from the previous study and the Extension study will be pooled for final analysis.

ELIGIBILITY:
Inclusion Criteria (NET-MED-002):

* Age ≥ 18 years

Inclusion Criteria (NET-MED-002-EXT):

* Age ≥ 18 years
* One (or more) chronic medical condition/s

Exclusion Criteria (NET-MED-002):

* Children under the age of 18 years
* Pregnant or lactating women - as confirmed by a home pregnancy test kit
* Current irregular heart rate (e.g. Atrial fibrillation) - as assessed by a targeted physical examination during screening
* Current shortness of breath, respiratory distress, or other clinical signs of hemodynamic instability - as assessed by a targeted physical examination during screening
* Prior major surgical and/or orthopedical and/or trauma in the thorax
* Participation in an investigational trial within 30 days of the screening visit
* Subjects that will not be able to complete the trial, according to the PI or SI evaluation

Exclusion Criteria (NET-MED-002-EXT)

* Children under the age of 18 years
* Prior major trauma in the thorax
* Participation in an investigational trial within 30 days of the screening visit
* Subjects that will not be able to complete the trial, according to the PI or SI evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females, 18 years old and above willing and able to provide an informed consent and eligible according to the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2021-02-21 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
Proportion of accurate spot HR while the Neteera 130H located behind the subject. | During 60 seconds, from t = 0:00 min to t = 1:00
  Proportion of accurate spot HR (BPM) measurements of the investigated device, while located behind the subject, in sitting position compared to the reference device measurements
Proportion of accurate spot RR while the Neteera 130H located behind the subject. | During 60 seconds, from t = 0:00 min to t = 1:00
  Proportion of accurate spot RR (BrPM) measurements of the investigated device in sitting position, while located behind the subject, compared to reference device (capnograph) measurements

SECONDARY OUTCOMES:
Repeating the primary endpoints in sitting position while the investigated device is located in front of the subject. | During 60 seconds, from t = 0:00 min to t = 1:00
  1) Repeating the primary endpoints in sitting position while the investigated device is located in front of the subject.
Repeating the previous endpoints (where applicable) in sleep posture/lying in bed position, while the investigated device is located above of the subject. | During 60 seconds
  Repeating the previous endpoints (where applicable) in sleep posture/lying in bed position, while the investigated device is located above of the subject.
Repeating previous endpoint positions (where applicable) comparing investigated device continuous HR and RR measurements to reference device continuous measurements | During 5 minutes of the continuous measurement
  Repeating previous endpoint positions (where applicable) comparing investigated device continuous HR and RR measurements to reference device continuous measurements

OTHER OUTCOMES:
Safety Endpoint | from screening until the end of study measurements
  Percent of subjects with device related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, MD, Principal Investigator — JBR Clinical Research
Locations (2):
- JBR Clinical Research, Millcreek, Utah, United States
- Shaare Zedek Medical Center, Jerusalem, Israel